CLINICAL TRIAL: NCT01568619
Title: Validation of Electrical Cardiometry Versus Fick Method to Measure Stroke Volume and Cardiac Output in Patients With or Suspected of Having Heart Failure
Brief Title: Validation of Electrical Cardiometry Versus Fick Method in Cardiac Output Measurement
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yandong Jiang, Assistant Professor, Massachusetts General Hospital
Other Study IDs: AESCULON
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Heart Failure
Keywords: cardiopulmonary exercise test; cardiac output
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators would like to find out if AESCULON®, a new device that non-invasively and continuously measures cardiac output using electrical cardiometry, works as well as one existing method--Fick method in patients undergoing cardiopulmonary exercise testing.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 yd;
* Level 3 cardiopulmonary exercise testing.

Exclusion Criteria:

* Proven or suspected disease involving severe aortic regurgitation;
* Implanted with a rate-responsive cardiac pacemaker;
* Pneumothorax or pleural effusion;
* Skin lesion(s) at the place where the electrode is supposed to be applied;
* Allergic to adhesive of ECG electrodes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of 18 years or older who undergo cardiopulmonary exercise testing (CPET) with invasive hemodynamic monitoring for their routine care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
difference in CO measurements with two methods | two weeks after finishing the exercise test
  the true difference between the two CO measurements is 10% of the mean CO

CONTACTS AND LOCATIONS:
Overall Officials: Yandong Jiang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States